CLINICAL TRIAL: NCT01518387
Title: Phase III Open Study of BAY 77 1931 (Lanthanum Carbonate) in Patients With Hyperphosphatemia Undergoing Continuous Ambulatory Peritoneal Dialysis (CAPD)
Brief Title: Open Study of BAY77-1931 (Lanthanum Carbonate) in Continuous Ambulatory Peritoneal Dialysis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11878
Record Dates: First submitted 2012-01-18; First posted 2012-01-26 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Hyperphosphatemia
Keywords: Hyperphosphatemia in ESRD (End Stage Renal Disease) patients on dialysis
MeSH Terms: conditions — Hyperphosphatemia; Kidney Failure, Chronic | interventions — lanthanum carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): 750-2250mg/day, tid, 8 weeks
  Interventions: Drug: Lanthanum Carbonate (BAY77-1931)

INTERVENTIONS:
Drug: Lanthanum Carbonate (BAY77-1931)

SUMMARY:
The purpose of this study is to assess the effect on reduction of serum phosphate and the safety of BAY77-1931 (lanthanum carbonate) in patients with hyperphosphatemia undergoing continuous ambulatory peritoneal dialysis.

ELIGIBILITY:
Inclusion Criteria:

* Serum phosphate levels: >5.0 mg/dL and <11.0 mg/dL 2 weeks after the initiation of the washout period
* Out-patient
* Undergoing CAPD for at least previous 3 consecutive months

Exclusion Criteria:

* Who may not enable to continue CAPD
* Serum phosphate levels of >=10.0 mg/dL at the start of the washout period or >=11.0 mg/dL 2 week after
* Corrected serum calcium level of <7.0 mg/dL at the start of the washout period or >=11.0 mg/dL 2 week after
* Serum intact PTH (Parathyroid) of >=1000 pg/mL at the start of the washout period
* Pregnant woman, or lactating mother
* Significant gastrointestinal disorders including known acute peptic ulcer
* Liver dysfunction
* History of cardiovascular or cerebrovascular diseases

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2006-01; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in serum phosphate levels at the end of the treatment period | Baseline to Week 8

SECONDARY OUTCOMES:
Number of participants achieving the target PSPL (Pre-dialysis serum phosphate level) and time to achievement | Week 8
Serum calcium level corrected by serum albumin level at the end of the treatment period | Week 8
Serum calcium x phosphate product at the end of the treatment period | Week 8
Serum intact-PTH (Parathyroid) levels at the end of the treatment period | Week 8
Safety variables will be summarized using descriptive statistics based on adverse events collection | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (11):
- Japan (11):
  - Fukuoka, Fukuoka
  - Gifu, Gifu
  - Hiroshima, Hiroshima
  - Asahikawa, Hokkaido
  - Kamakura, Kanagawa
  - Yokosuka, Kanagawa
  - Ōsaki, Miyagi
  - Sendai, Miyagi
  - Okayama, Okayama-ken
  - Tokushima, Tokushima
  - Meguro-ku, Tokyo